CLINICAL TRIAL: NCT05241080
Title: Covid -19 Related Stress Among Final Year BAMS Students During Lock Down Days in Kerala-A Cross Sectional Study
Brief Title: Stress Among Final Year BAMS Students in Relation With Covid Lockdown Through CSSQ-a Cross Sectional Survey
Status: Completed | Type: Observational
Sponsor: Amrita Vishwa Vidyapeetham (Other)
Collaborators: Amrita Viswa Vidyapeetham (Unknown)
Responsible Party: Principal Investigator, Dr.Preethi Mohan, Associate professor, Amrita Vishwa Vidyapeetham
Other Study IDs: Not yet assaigned
Record Dates: First submitted 2022-02-14; First posted 2022-02-15 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: Covid Related Psychological Stress
Keywords: Stress,covid,lock down days
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Survey — It is a survey based on questionnaire

SUMMARY:
We were randomly selected the ayurveda colleges in Kerala.Selected final year BAMS students as participants.we have also selected a group of 5 members for data colle tion.we have selected a validated Covid stress questionnaire and circulated through what's app and Gmail.we were received responses from each college with .we analyzed and interpreted data.

DETAILED DESCRIPTION:
We were randomly selected the ayurveda colleges in Kerala.Selected final year BAMS students as participants.we have also selected a group of 5 members for data colle tion.we have selected a validated Covid stress questionnaire and circulated through what's app and Gmail.we were received responses from each college with .we analyzed and interpreted data.

ELIGIBILITY:
Inclusion Criteria 1.final year BAMS 2.irrespective of gender

-

Exclusion Criteria:

* age group other than 20-22 yrs

Ages: 20 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: All final year students Of BAMS studying inside Kerala.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2021-11-30 (Actual); Primary Completion 2021-12-10 (Actual); Study Completion 2021-12-10 (Actual)

PRIMARY OUTCOMES:
Likert scale | 10 days
  4 point likert scale questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Dr.preethi Mohan, BAMS MD, Principal Investigator — Amrita Viswa Vidyapeetham; Delvin T Robin, Principal Investigator — Amrita Vishwa Vidyapeetham
Locations (1):
- Dr Preeti, Kollam, Kerala, India

IPD SHARING:
Plan to Share IPD: No